CLINICAL TRIAL: NCT06657183
Title: Enhanced Care Management (ECM) and Continuous Monitoring of Vital Signs With Alio Smart Patch Wearable Sensor in Adult Cancer Patients Receiving Chemotherapy With Moderate or High Risk of Febrile Neutropenia or Immunotherapy
Brief Title: ECM and Monitoring w/ Alio Smart Patch in Cancer Pts Receiving Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4124
Record Dates: First submitted 2024-10-17; First posted 2024-10-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Febrile Neutropenia
Keywords: Alio Smart Patch
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Remote Monitoring with Smartpatch (Experimental): Participants will be continuously monitored through the device, providing crucial physiological data. The Smartpatch will allow for early detection of chemotherapy-related toxicities.
  Interventions: Device: Alio Smart Patch™

INTERVENTIONS:
Device: Alio Smart Patch™ — Alio Smart Patch is a non-invasive wearable biosensor that combines a unique, multi-sensor, wearable device with a provided- based portal to track sequentially the participant's physiologic, hematologic and electrolyte data. It works in conjunction with a home hub data relay system and an end-to-end cloud software data path. The system has been developed to enable home monitoring for multiple key metrics by healthcare provider caring for participants.
  Enhanced Care Management (ECM) is a comprehensive, system-centric approach crafted to bridge the latent gaps in traditional care paradigms. ECM provides an exhaustive review of a participant's medical history and their personalized social needs, addressing both in a cohesive, participant-focused strategy.
  This intervention couples Quantify Remote Care's Enhanced Care Management with the Alio Smart Patch technology.

SUMMARY:
Undergoing cancer treatment comes with various risks and side effects. This clinical trial aims to reduce those risks and side effects through continuous monitoring of vital signs and blood levels. The goal is to see if potential side effects can be identified and treated sooner.

During this study, participants will wear an Alio Smartpatch™. The Alio Smartpatch™ is a wireless remote monitoring system. This device will measure participants' vital signs and blood levels. Participants will also be asked to use continuous glucose monitors to measure their glucose levels. The data collected on each participant from these devices will be remotely monitored at all times by clinical staff at a company known as Quantify Remote Care. If a participant's results look like they are experiencing a side effect, the participant will be contacted immediately by Quantify Remote Care team. The Quantify Remote Care team will function as an extension of the participant's cancer clinical team and will relay any significant issues back to them. Quantify Health also provides dietary and mental health support as needed for all participants.

DETAILED DESCRIPTION:
Cancer care often involves aggressive treatments like chemotherapy, exposing patients to serious risks, such as febrile neutropenia, and other chemotherapy-related complications. Current care models depend heavily on patients reporting issues, often leading to delays in necessary intervention. This emphasizes the need for a more proactive and sophisticated approach to patient monitoring and care management. Modern wearable devices provide continuous objective data with the goal of enhancing cancer care. Patient-generated health data (PGHD), or health-related data gathered from patients to help address a health concern, are used increasingly in oncology to make regulatory decisions and evaluate quality of care. PGHD include self-reported health and treatment histories and patient-reported outcomes (PROs). A recent prospective study assessed the feasibility of monitoring of physical activity using a commercial wearable device and collecting electronic patient-reported outcomes (ePROs) during radiotherapy (RT) for head and neck cancer (HNC). In this study 29 patients were enrolled; step data were recorded on 70% of the days during patients' RT courses, and there were only 11 patients (38%) for whom step data were collected on at least 80% of days during RT. feasibility end point was not achieved suggesting that rigorous workflows are required to achieve continuous activity monitoring during RT. However, the findings are consistent with previous reports indicating that wearable device data can help identify patients who are at risk for unplanned hospitalization. In another study, patients with early stage breast cancer were enrolled prior to starting chemotherapy. Patients received a Fitbit Charge HR and were instructed to wear it and sync at least weekly throughout chemotherapy and up to six months post therapy. Patients completed baseline surveys, and treatment information was collected from their medical records. Fitbit data was downloaded from the Fitabase data management platform. To assess utility, they evaluated how many days patients wore their Fitbit for at least 10 hours. Fitbit use during breast cancer chemotherapy was poor in the absence of prompts to encourage wear. Interventions including phone calls, texts, to maintain adherence are likely necessary to increase wear in active treatment settings. Cancer patients receiving chemotherapy who are at high risk of febrile neutropenia, infections or complications in general, would benefit from a new remote monitoring model that not only monitors data but records, trends and delivers actionable clinical insights regarding the patient status with a goal of intervening early and evaluate potential toxicities and complications from treatment. The goal would be to assess compliance in addition to decrease frequency of emergency department visits as well as unplanned hospital admissions.

Quantify Remote Care's Enhanced Care Management (ECM) program aims to proactively manage patients undergoing complex treatment regimens, particularly those at high risk for complications. Our ECM program harnesses cutting-edge technology to enable continuous, real-time monitoring of a variety of physiological metrics, allowing for immediate intervention at the earliest signs of patient distress. One such technology is the Alio Smart Patch, originally developed for monitoring patients with end-stage renal disease undergoing hemodialysis. The wearable biosensor offers multi-sensor capabilities, capturing physiologic, hematologic, and electrolyte data in real time. This data is then channeled into a provider-based portal for seamless integration into clinical decision-making processes.

This pilot study aims to evaluate the efficacy of Quantify Remote Care's ECM program in cancer patients receiving chemotherapy, who are notably at higher risk of complications from treatment. Participants will be equipped with the Alio Smart Patch, giving healthcare providers 24-hour access to essential medical data, thereby enabling timely interventions to prevent severe complications.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following inclusion criteria in order to be eligible to participate in the study:
* Subjects have a diagnosis of soft tissue sarcoma, NSCLC, HNSCC, breast, pancreatic cancer, or melanoma
* For Cohort 1 (n=15), participants are eligible if starting on a new chemotherapy regimen with either: (i) high risk (> 20%) of febrile neutropenia as per NCCN MGF guidelines; or (ii) intermediate risk for febrile neutropenia AND one or more risk factors for febrile neutropenia:

  * Age > or equal to 65 years
  * Advanced disease
  * Previous Chemotherapy or Radiation therapy
  * Preexisting neutropenia or bone marrow involvement with tumor
  * Infection
  * Open wounds or surgery in last 4 weeks
  * Poor performance status or poor nutritional status
  * Poor renal function (cr clearance <50)
  * Total Bilirubin >1.5 upper limit of normal
  * Cardiovascular Disease
  * Multiple Co-morbidities
  * HIV infection
  * BMI > 2.0
* For Cohort 2 (n=15) participants are eligible if starting on immunotherapy alone, or concurrent chemo-immunotherapy.
* Participants are capable of giving informed consent
* Participants must be able to read and/or to speak English
* Participants who are 18 years of age or older
* Expected chemotherapy treatment duration of at least 12 weeks

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * Participants who cannot read or speak English
  * Participants without any cellphone access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Participant compliance | Up to 12 weeks from entering study
  Rate of participant compliance will be measured. Alio Smartpatch Compliance is defined as >=80% daily use, reflecting participant adherence to the prescribed monitoring regimen.

SECONDARY OUTCOMES:
Identification of febrile neutropenia symptoms | Up to 13 weeks from entering study
  Success rate of Alio Smart Patch under QRC ECM ability to identify febrile neutropenia symptoms.
Participant satisfaction: Usability | Up to 13 weeks from entering study
  The average participant satisfaction score will be measured by assessing participant satisfaction concerning the usability of Alio Smart Patch under QRC ECM.
Participant satisfaction: Comfort | Up to 13 weeks from entering study
  The average participant satisfaction score will be measured by assessing participant satisfaction concerning the comfort of using Alio Smart Patch under QRC ECM.
Participant satisfaction: Overall Experience | Up to 13 weeks from entering study
  The average participant satisfaction score will be measured by assessing participant satisfaction concerning the overall experience of using Alio Smart Patch under QRC ECM.
Clinical effectiveness of the integrated QRC ECM and smartpatch as measured by frequency of emergency care | Up to 13 weeks from entering study
  To validate the clinical effectiveness of the QRC ECM with smartpatch method, metrics will include the number of emergency room visits to determine if there is a reduction.
Clinical effectiveness of the integrated QRC ECM and smartpatch as measured by early detection | Up to 13 weeks from entering study
  To validate the clinical effectiveness of the QRC ECM with smartpatch method, metrics will include the rate of early detection.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Montero, MD, MBA, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals Seidman Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, University Hospitals Cleveland Medical Center Seidman Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study